CLINICAL TRIAL: NCT04785573
Title: The Effect of Mastiha Oil in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Associate Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mastiha_oil_GR_477
Record Dates: First submitted 2021-02-16; First posted 2021-03-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — mastiha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants with metabolic disorders will be subjected to nutritional counsel and the intake of 1 soft gel capsule daily for a total of 3 months.
  Interventions: Dietary Supplement: Mastiha oil
- Control group (No Intervention): Participants with metabolic disorders will be subjected to nutritional counsel for a total of 3 months.

INTERVENTIONS:
Dietary Supplement: Mastiha oil — 1 soft gel capsule of Mastiha oil every day for 3 months
  Arms: Intervention group

SUMMARY:
Mastiha Oil is a 100% natural product of the Mediterranean, extracted from the resin of Mastiha. Over 90 compounds have been identified in Mastiha oil, with monoterpenes exhibiting favorable effects in regulating mechanisms of oxidative stress and inflammation. The aim of this study is to determine the effect of Mastiha oil in adults with Metabolic Syndrome. 90 participants will be allocated to two groups, (45 in intervention group and 45 in control group). Mastiha oil will be provided in the form of soft gel capsules to the intervention group, whereas the control group will not consume the capsules. Both groups will receive standard nutritional counselling. The intervention will last 3 months.

The effects of the intervention will be evaluated via clinical and laboratory markers.

ELIGIBILITY:
Inclusion Criteria:

* 30 years < Age < 75 years
* Metabolic Syndrome cardiometabolic parameters
* A stable weight for ≥ 3 months pre-intervention
* An unchanged treatment regimen for ≥ 6 months pre-intervention

Exclusion Criteria:

* Hepatotoxic Medication
* Untreated Diabetes Mellitus
* Dysthyroidism, hypopituitarism, Cushing syndrome / disease
* Pregnancy, lactation
* Psychiatric or mental disorder
* Any use of antioxidant-phytochemical rich supplement, vitamin D supplement, anti-, pre- or pro-biotics within 3 months pre-intervention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change in blood total cholesterol | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in insulin sensitivity | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in blood triglycerides | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in blood LDL | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups

SECONDARY OUTCOMES:
Change in blood CRP | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in blood MPO | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in blood IL-6 | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups
Change in blood antioxidant potential | 3 months
  Levels will be evaluated pre and prost intervention in both control and intervention groups

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Harokopio University, Athens, Attica
  - Andriana Kaliora, Athens

REFERENCES:
- [Derived] Gioxari A, Amerikanou C, Valsamidou E, Kleftaki SA, Tzavara C, Kalaitzopoulou A, Stergiou I, Smyrnioudis I, Kaliora AC. Chios mastiha essential oil exhibits antihypertensive, hypolipidemic and anti-obesity effects in metabolically unhealthy adults - a randomized controlled trial. Pharmacol Res. 2023 Aug;194:106821. doi: 10.1016/j.phrs.2023.106821. Epub 2023 Jun 15. PMID 37329633